CLINICAL TRIAL: NCT04909411
Title: Consequences of a Maternal-fetal Chikungunya Virus Infection. Neurocognitive and Sensory Assessment Around the Age of 13.
Brief Title: Consequences of a Maternal-fetal Chikungunya Virus Infection
Acronym: CHIK13+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/CHU/07
Record Dates: First submitted 2021-05-28; First posted 2021-06-01 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Chikungunya Virus Infection
MeSH Terms: conditions — Chikungunya Fever | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposed arm (Other): child infected with chikungunya virus during childbirth
  Interventions: Other: OPHTHALMOLOGICAL ASSESSMENT; Other: NEUROPSYCHOLOGICAL ASSESSMENT
- Non-exposed arm (Other): child not infected with the chikungunya virus at the time of childbirth, verifying the matching criteria specified
  Interventions: Other: OPHTHALMOLOGICAL ASSESSMENT; Other: NEUROPSYCHOLOGICAL ASSESSMENT

INTERVENTIONS:
Other: OPHTHALMOLOGICAL ASSESSMENT — assessment of eye mobility (search for heterophoria or strabismus), visual acuity, visual fields, external structures and funduscopic examination
Other: NEUROPSYCHOLOGICAL ASSESSMENT — completion of WISC-5, Vineland Adaptive Behavior Scale II and Strengths and Difficulties Questionnaire

SUMMARY:
Chikungunya is an infectious disease caused by an alphavirus transmitted by the Aedes mosquitoes which has known a worldwide expansion since its re-emergence in 2004. Regarding to an unprecedented epidemic, Reunionese pediatricians described in 2005-2006 a vertical maternal-fetal transmission of this virus, at the time of childbirth. Since then, this mode of transmission has been widely confirmed, with an absolute risk estimated between 15.5% and 48.3%. The main consequences for the child are neuromotor, neurosensory or neurocognitive. They were studied around the age of 2 in 33 children in the CHIMERE cohort, as well as at the age of 5 in a small fraction of these children followed at the C.A.M.S.P (Center for Early Medico-Social Action). The results suggested an overall delay in psychomotor acquisitions secondary to neonatal infection, affecting the functions of the prefrontal region (in particular coordination and language). Performance was correlated with the severity of the clinical presentation (more severe in case of encephalitis or encephalopathy) while remaining suboptimal in children with uncomplicated infection. During neurodevelopmental monitoring, other disturbing traits complemented the spectrum of problems presented by these children, such as microcephaly, cerebral palsy, epilepsy, interaction disorder or attention deficit disorder. At around age 10, the investigators reassessed 21 of these children using the Childhood Cognitive Function and Learning (EDA) screening test. The investigators would now like to confirm and characterize their impairments using a battery of confirmatory tests around the age of 13.

ELIGIBILITY:
Inclusion Criteria:

* Child born between March 2005 and July 2006
* Of which the mother identified in the CHIMERE cohort or the perinatal register of maternities
* Exposed: child infected with the chikungunya virus at the time of childbirth
* Not exposed: child not infected with the chikungunya virus at the time of childbirth, verifying the matching criteria specified in chapter 5.2
* Affiliated to a social insurance

Exclusion Criteria:

* Prematurity <33 weeks
* Prenatal alcoholization authenticated by fetal alcohol syndrome
* Intellectual disability or secondary epilepsy of origin other than CHIKV infection (caused by ACSOS or any other cause of brain damage of inflammatory, metabolic or infectious origin)

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Total intelligence quotient | Month 3 (+/- 1 month)
  Evaluation of total intelligence quotient with Wechsler Intelligence Scale for Children-5

CONTACTS AND LOCATIONS:
Overall Officials: Raphaelle SARTON, MD, Principal Investigator — CHU de La Réunion
Locations (1):
- CHU de La Réunion, Saint-Pierre, Reunion